CLINICAL TRIAL: NCT00107952
Title: A Phase 3, Randomized, Double-Blind, Parallel-Group, Multinational Trial of Intravenous Telavancin Versus Vancomycin for Treatment of Hospital-Acquired Pneumonia With a Focus on Patients With Infections Due to Methicillin-Resistant Staphylococcus Aureus
Brief Title: Comparison of Telavancin and Vancomycin for Hospital-acquired Pneumonia Due to Methicillin-resistant Staphylococcus Aureus
Acronym: ATTAIN1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Steven Barriere, Pharm.D., Vice President, Clinical and Medical Affairs, Theravance, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0015
Record Dates: First submitted 2005-04-11; First posted 2005-04-12 (Estimated); Results first posted 2009-12-08 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Bacterial Pneumonia
Keywords: Nosocomial pneumonia; MRSA
MeSH Terms: conditions — Pneumonia, Bacterial; Healthcare-Associated Pneumonia | interventions — telavancin; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telavancin (Experimental)
  Interventions: Drug: Telavancin
- Vancomycin (Active Comparator)
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Telavancin — Telavancin 10 mg/kg/day IV for up to 21 days.
  Other Names: TD-6424; VIBATIV
  Arms: Telavancin
Drug: Vancomycin — Vancomycin 1 Gm IV q 12 hrs for up to 21 days
  Arms: Vancomycin

SUMMARY:
Study 0015 (NCT00107952) compares the safety and effectiveness of an investigational drug, telavancin, with vancomycin for the treatment of hospital-acquired pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Clinical signs and symptoms consistent with pneumonia acquired after at least 48 hours of continuous stay in an inpatient acute or chronic care facility or acquired within 7 days after being discharged from a hospitalization of greater than or equal to 3 days duration.

Exclusion Criteria:

* Received more than 24 hours of potentially effective systemic (IV, IM or PO) antibiotic therapy for Gram-positive pneumonia immediately prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 761 (Actual)
Dates: Start 2005-02; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: G. Ralph Corey, MD, Principal Investigator — Duke University
Locations (1):
- Baystate Medical Center, Springfield, Massachusetts, United States

REFERENCES:
- [Derived] McKinnell JA, Corman S, Patel D, Leung GH, Gordon LM, Lodise TP. Effective Antimicrobial Stewardship Strategies for Cost-effective Utilization of Telavancin for the Treatment of Patients With Hospital-acquired Bacterial Pneumonia Caused by Staphylococcus aureus. Clin Ther. 2018 Mar;40(3):406-414.e2. doi: 10.1016/j.clinthera.2018.01.010. Epub 2018 Feb 15. PMID 29454592
- [Derived] Smart JI, Corey GR, Stryjewski ME, Wang W, Barriere SL. Assessment of Minimum Inhibitory Concentrations of Telavancin by Revised Broth Microdilution Method in Phase 3 Hospital-Acquired Pneumonia/Ventilator-Associated Pneumonia Clinical Isolates. Infect Dis Ther. 2016 Dec;5(4):535-544. doi: 10.1007/s40121-016-0133-y. Epub 2016 Oct 7. PMID 27718118
- [Derived] Barriere SL, Stryjewski ME, Corey GR, Genter FC, Rubinstein E. Effect of vancomycin serum trough levels on outcomes in patients with nosocomial pneumonia due to Staphylococcus aureus: a retrospective, post hoc, subgroup analysis of the Phase 3 ATTAIN studies. BMC Infect Dis. 2014 Apr 4;14:183. doi: 10.1186/1471-2334-14-183. PMID 24708675

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment Period: 08Feb05 to 11Jul07
Groups:
- Telavancin: Patients with Gram-positive hospital acquired pneumonia (HAP) (primarily due to MRSA) were randomized to receive telavancin 10 mg/kg IV every 24 hrs.
- Vancomycin: Patients with Gram-positive hospital acquired pneumonia (HAP)(primarily due to MRSA) were randomized to receive vancomycin 1 Gm IV administered every 12 hrs.
Period: Overall Study
Arm/Group | Telavancin | Vancomycin
Started | 381 | 380
Completed | 286 | 299
Not Completed | 95 | 81
Not completed — Death | 75 | 61
Not completed — Lost to Follow-up | 0 | 3
Not completed — Withdrawal by Subject | 9 | 6
Not completed — Other | 2 | 5
Not completed — Never received study treatment | 9 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telavancin | Vancomycin | Total
Number analyzed (Participants) | 372 | 374 | 746
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 170 | 162 | 332
  >=65 years | 202 | 212 | 414
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (19.2) | 64 (17.3) | 64 (18.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137 | 161 | 298
  Male | 235 | 213 | 448
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 78 | 66 | 144
  Not Hispanic or Latino | 294 | 308 | 602
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 91 | 87 | 178
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 10 | 14 | 24
  White | 267 | 272 | 539
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Argentina | 24 | 24 | 48
  Australia | 20 | 25 | 45
  Belgium | 3 | 5 | 8
  Brazil | 12 | 14 | 26
  Canada | 14 | 10 | 24
  Chile | 9 | 5 | 14
  Croatia | 28 | 31 | 59
  Czech Republic | 0 | 1 | 1
  France | 15 | 17 | 32
  Greece | 4 | 8 | 12
  India | 44 | 41 | 85
  Israel | 25 | 24 | 49
  Italy | 3 | 4 | 7
  Malaysia | 13 | 7 | 20
  Malta | 2 | 1 | 3
  Peru | 2 | 3 | 5
  Poland | 0 | 2 | 2
  South Africa | 2 | 2 | 4
  Taiwan | 29 | 34 | 63
  Turkey | 2 | 1 | 3
  United Kingdom | 4 | 2 | 6
  United States | 117 | 113 | 230
Diabetes Status [Number; unit: Participants]
  Diabetic | 100 | 100 | 200
  Non-Diabetic | 272 | 274 | 546
History of Pneumonia [Number; unit: participants]
  Prior history of pneumonia | 62 | 53 | 115
  No prior history of pneumonia | 310 | 321 | 631
Ventilator Status [Number; unit: Participants]
  Ventilated | 170 | 171 | 341
  Non-ventilated | 202 | 203 | 405

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response
Description: Clinical Response: Categorical (Cured, Failed or Indeterminate)
  * Failure is at least one of the following: Persistence or progression of signs and symptoms of pneumonia that still require antibiotic therapy; Termination of study med due to "lack of efficacy"; Death on or after Day 3 attributable to primary infection
  * Cure: Signs and symptoms of pneumonia improved to the point that no further antibiotics for pneumonia were required, and baseline radiographic findings improved or did not progress.
  * Indeterminate: Inability to determine outcome
Time Frame: 7 - 14 days following end of antibiotic treatment
Measure: Number; unit: participants
Arm/Group | Telavancin | Vancomycin
Number analyzed (Participants) | 372 | 374
participants
  Cured | 214 | 221
  Failure | 46 | 68
  Indeterminate | 56 | 41
  Missing | 56 | 44
Statistical Analysis 1: Comparison: Telavancin vs Vancomycin; Test type: Non-Inferiority or Equivalence — Non-inferiority margin of 20% was specified based on historical regulatory precedent; p-values were not calculated in deference to confidence intervals; Risk Difference (RD) = -1.6, 95% CI [-8.6 to 5.5] — Statistical analysis applies to "cure"

ADVERSE EVENTS:
Arm/Group | Telavancin | Vancomycin
Serious Adverse Events (participants affected / at risk) | 127/372 | 88/374
Other Adverse Events (participants affected / at risk) | 321/372 | 317/374
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telavancin (N=372) | Vancomycin (N=374)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Acute Coronary Syndrome (Cardiac disorders) | 1 | 0
Angina Unstable (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 3
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 2 | 1
Cardiac Arrest (Cardiac disorders) | 2 | 4
Cardiac failure (Cardiac disorders) | 1 | 2
Cardiac failure congestive (Cardiac disorders) | 4 | 3
Cardio-Respiratory Arrest (Cardiac disorders) | 1 | 0
Cardiogenic Shock (Cardiac disorders) | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 1
Left Ventricular Failure (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 1 | 1
Myocardial Ischaemia (Cardiac disorders) | 2 | 1
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 2
Ventricular tachycardia (Cardiac disorders) | 1 | 3
Pituitary Haemorrhage (Endocrine disorders) | 1 | 0
Duodenal perforation (Gastrointestinal disorders) | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 | 2
Haematemesis (Gastrointestinal disorders) | 0 | 1
Oesophagitis ulcerative (Gastrointestinal disorders) | 1 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 1
Peritonitis (Gastrointestinal disorders) | 1 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 | 1
Death (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Multi-organ Failure (General disorders) | 11 | 8
Sudden Cardiac Death (General disorders) | 0 | 1
Hepatic Failure (Hepatobiliary disorders) | 0 | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 1 | 0
Abdominal Sepsis (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0
Catheter sepsis (Infections and infestations) | 0 | 1
Clostridium Colitis (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Mediastinitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 6 | 8
Pyelonephritis chronic (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 6 | 4
Septic shock (Infections and infestations) | 13 | 13
Urinary Tract Infection (Infections and infestations) | 0 | 1
Urinary Tract Infection Bacterial (Infections and infestations) | 0 | 1
Urosepsis (Renal and urinary disorders) | 2 | 0
Injury asphyxiation (Injury, poisoning and procedural complications) | 0 | 1
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Blood creatinine increased (Investigations) | 3 | 0
Diabetic hyperosmolar non-ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Fluid Overload (Metabolism and nutrition disorders) | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hepatic Neoplasm Malignant (Nervous system disorders) | 1 | 0
Cerebral Haemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular Infarction (Nervous system disorders) | 2 | 0
Cerebrovascular Accident (Nervous system disorders) | 2 | 2
Convulsion (Nervous system disorders) | 0 | 2
Encephalopathy (Nervous system disorders) | 1 | 0
Haemorrhage Intracranial (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Hypoxic encephalopathy (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Nervous System Disorder (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0
Status epilepticus (Nervous system disorders) | 1 | 0
Anuria (Renal and urinary disorders) | 1 | 0
Obstructive Uropathy (Renal and urinary disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 11 | 3
Renal Insufficiency (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic Obstructive Airways Disease Exacerbated (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dependence on Respirator (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 14 | 11
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Subcutaneous Emphysema (Skin and subcutaneous tissue disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
Gangrene (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0
Poor peripheral circulation (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 3 | 2
Shock Haemorrhagic (Vascular disorders) | 3 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Telavancin (N=372) | Vancomycin (N=374)
Anemia (Blood and lymphatic system disorders) | 30 | 49
Thrombocythaemia (Blood and lymphatic system disorders) | 7 | 1
Atrial fibrillation (Cardiac disorders) | 16 | 18
Bradycardia (Cardiac disorders) | 6 | 10
Cardiac failure congestive (Cardiac disorders) | 10 | 12
Tachycardia (Cardiac disorders) | 5 | 9
Abdominal Distension (Gastrointestinal disorders) | 6 | 2
Abdominal Pain (Gastrointestinal disorders) | 4 | 9
Constipation (Gastrointestinal disorders) | 32 | 36
Diarrhoea (Gastrointestinal disorders) | 47 | 54
Dyspepsia (Gastrointestinal disorders) | 3 | 6
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 7 | 8
Nausea (Gastrointestinal disorders) | 27 | 19
Vomiting (Gastrointestinal disorders) | 21 | 19
Anasarca (General disorders) | 6 | 8
Infusion site phlebitis (General disorders) | 6 | 5
Multi-organ Failure (General disorders) | 12 | 8
Non-Cardiac Chest Pain (General disorders) | 8 | 7
Oedema Peripheral (General disorders) | 20 | 26
Pain (General disorders) | 8 | 7
Bacteraemia (Infections and infestations) | 5 | 8
Oral Candidiasis (Infections and infestations) | 9 | 5
Pneumonia (Infections and infestations) | 8 | 8
Sepsis (Infections and infestations) | 9 | 10
Septic shock (Infections and infestations) | 15 | 13
Urinary Tract Infection (Infections and infestations) | 19 | 21
Excoriation (Injury, poisoning and procedural complications) | 7 | 8
Alanine Aminotransferase increased (Investigations) | 7 | 9
Aspartate Aminotransferase increased (Investigations) | 6 | 8
Blood Alkaline Phosphatase Increased (Investigations) | 7 | 5
Blood Creatinine Increased (Investigations) | 11 | 6
Electrocardiogram QT Corrected interval prolonged (Investigations) | 6 | 2
Fluid Overland (Metabolism and nutrition disorders) | 10 | 9
Hyperglycaemia (Metabolism and nutrition disorders) | 10 | 11
Hyperkalaemia (Metabolism and nutrition disorders) | 11 | 9
Hypoalbuminaemia (Metabolism and nutrition disorders) | 11 | 16
Hypocalcaemia (Metabolism and nutrition disorders) | 6 | 6
Hypoglycaemia (Metabolism and nutrition disorders) | 12 | 9
Hypokalemia (Metabolism and nutrition disorders) | 30 | 41
Hypomagnesaemia (Metabolism and nutrition disorders) | 7 | 16
Hyponatremia (Metabolism and nutrition disorders) | 8 | 11
Malnutrition (Metabolism and nutrition disorders) | 6 | 3
Metabolic acidosis (Metabolism and nutrition disorders) | 8 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 6
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 5 | 6
Headache (Nervous system disorders) | 10 | 13
Agitation (Psychiatric disorders) | 10 | 12
Anxiety (Psychiatric disorders) | 10 | 20
Depression (Psychiatric disorders) | 4 | 7
Insomnia (Psychiatric disorders) | 16 | 32
Haematuria (Renal and urinary disorders) | 8 | 7
Renal Failure Acute (Renal and urinary disorders) | 18 | 10
Renal Insufficiency (Renal and urinary disorders) | 5 | 8
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 8
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 16 | 15
Decubitis Ulcer (Skin and subcutaneous tissue disorders) | 22 | 26
Erythema (Skin and subcutaneous tissue disorders) | 7 | 6
Rash (Skin and subcutaneous tissue disorders) | 21 | 10
Hypertension (Vascular disorders) | 11 | 14
Hypotension (Vascular disorders) | 23 | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less